CLINICAL TRIAL: NCT00960687
Title: A Single-Dose, Bioequivalence Study of 105 mg Fenofibric Acid Tablets Versus 145 mg TriCor® (Fenofibrate) Tablets Under Fed Conditions(Standard Meal)
Brief Title: Fed Bioequivalence Study of Fenofibric Acid Versus TriCor® (Fenofibrate)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-028-07-1008; R07-1033
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Results first posted 2009-10-14 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: healthy; pharmacokinetics; therapeutic equivalency
MeSH Terms: interventions — fenofibric acid; Fenofibrate; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenofibric Acid (Fibricor™) (Experimental): 1 x 105 mg fenofibric acid (Fibricor™)tablet administered 30 minutes after the initiation of a standard breakfast.
  Interventions: Drug: Fenofibric Acid (Fibricor™) 105 mg Tablet
- Fenofibrate (Tricor®) (Experimental): 1 x 145 mg fenofibrate (Tricor®) tablet administered 30 minutes after the initiation of a standard breakfast.
  Interventions: Drug: Fenofibrate (Tricor®) 145 mg Tablet

INTERVENTIONS:
Drug: Fenofibric Acid (Fibricor™) 105 mg Tablet — 1 x 105 mg fenofibric acid (Fibricor™) tablet administered 30 minutes after the initiation of a standard breakfast.
  Other Names: Fibricor™
  Arms: Fenofibric Acid (Fibricor™)
Drug: Fenofibrate (Tricor®) 145 mg Tablet — 1 x 145 mg Fenofibrate (Tricor®) tablet administered 30 minutes after the start of a standard breakfast.
  Other Names: Tricor®
  Arms: Fenofibrate (Tricor®)

SUMMARY:
This study will evaluate the bioequivalence of 105 mg fenofibric acid tablets relative to 145 mg fenofibrate tablets in healthy volunteers when administered following a breakfast of standard composition. Safety and tolerability of this regimen will also be evaluated.

DETAILED DESCRIPTION:
Fenofibrate is rapidly and completely hydrolyzed to fenofibric acid, the active moiety. The primary objective of this study is to evaluate the bioequivalence of 105 mg fenofibric acid tablets relative to 145 mg fenofibrate tablets in healthy volunteers when administered following a breakfast of standard composition. Additionally, the safety and tolerability of this dosing regimen will be evaluated. Fifty-four healthy, non-smoking, non-obese, 18-45 year old, male and female volunteers will be randomly assigned in a crossover fashion to receive each of two dosing regimens (fenofibric acid and fenofibrate) in sequence with a 7 day washout period between dosing periods. On the morning of Day 1, subjects will receive either a single oral dose of the test formulation, fenofibric acid (1 x 105 mg tablet) or a single oral dose of the reference formulation, fenofibrate (1 x 145 mg tablet) 30 minutes after the initiation of a standard breakfast. After a 7 day washout period, on the morning of Day 8, subjects will receive the alternate regimen 30 minutes after the initiation of a standard breakfast. Fasting will continue for 4 hours after each dose. Blood samples will be drawn from all participants before dosing and for 72 hours post dose at times sufficient to adequately define the pharmacokinetics of fenofibric acid. Subjects will be monitored throughout their participation for adverse reactions to the study drug and/or procedures. Seated blood pressure and pulse will be measured prior to each dose and approximately 2 hours post-dose. All adverse experiences, whether elicited by query, spontaneously reported, or observed by clinic staff, will be documented in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age
* Non-smoking
* Non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures)
* Body mass index (BMI) less than 30
* Medically healthy on the basis of medical history and physical examination
* Hemoglobin > or = to 12g/dL
* Completion of the screening process within 28 days prior to dosing
* Provision of voluntary written informed consent

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to fenofibrate (fenofibric acid)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm. D., Principal Investigator — PRACS Institute

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-Four (54) non-obese, non-smoking, healthy adult volunteers, consisting of members of the community-at-large, were enrolled.
Pre-assignment Details: Ninety-nine (99) subjects were screened. Forty-five (45) subjects were screen failures. The remaining fifty-four subjects were enrolled, 47 of whom completed the study.
Groups:
- Fenofibric Acid 105 mg Tablets Then Fenofibrate 145 mg Tablets: On the morning of Day 1 subjects received one tablet of the test formulation, fenofibric acid 105 mg, 30 minutes after the initiation of a standard breakfast, followed by a 7 day washout period. On the morning of Day 8 subjects received one tablet of the reference formulation, fenofibrate 145 mg, 30 minutes after the initiation of a standard breakfast.
- Fenofibrate 145 mg Tablets Then Fenofibric Acid 105 mg Tablets: On the morning of Day 1 subjects received one tablet of the reference formulation, fenofibrate 145 mg, 30 minutes after the initiation of a standard breakfast, followed by a 7 day washout period. On the morning of Day 8 subjects received one tablet of the test formulation, fenofibric acid 105 mg, 30 minutes after the initiation of a standard breakfast.
Period: First Intervention
Arm/Group | Fenofibric Acid 105 mg Tablets Then Fenofibrate 145 mg Tablets | Fenofibrate 145 mg Tablets Then Fenofibric Acid 105 mg Tablets
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Fenofibric Acid 105 mg Tablets Then Fenofibrate 145 mg Tablets | Fenofibrate 145 mg Tablets Then Fenofibric Acid 105 mg Tablets
Started | 27 | 27
Completed | 23 (three subjects withdrew due to adverse events and one subject withdrew for personal reasons.) | 24 (two subjects withdrew due to adverse events and one subject withdrew for personal reasons.)
Not Completed | 4 | 3
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention
Arm/Group | Fenofibric Acid 105 mg Tablets Then Fenofibrate 145 mg Tablets | Fenofibrate 145 mg Tablets Then Fenofibric Acid 105 mg Tablets
Started | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fenofibric Acid 105 mg Tablets and Fenofibrate 145 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either fenofibric acid 105 mg or fenofibrate 145 mg, 30 minutes after the initiation of a standard meal.
Arm/Group | Fenofibric Acid 105 mg Tablets and Fenofibrate 145 mg Tablets
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours after drug administration.
Population: Pharmacokinetic analyses are based on 47 out of 54 enrolled subjects who completed this study.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fenofibric Acid 105 mg Tablets: Each subject received one tablet of fenofibric acid 105mg 30 minutes after the initiation of a standard breakfast.
- Fenofibrate 145 mg Tablets: Each subject received one tablet of fenofibrate 145mg 30 minutes after the initiation of a standard breakfast.
Arm/Group | Fenofibric Acid 105 mg Tablets | Fenofibrate 145 mg Tablets
Number analyzed (Participants) | 47 | 47
ng/mL | 8,545.50 (1,792.62) | 9,456.66 (1,741.55)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: Pharmacokinetic analyses are based on 47 out of 54 enrolled subjects who completed this study.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Fenofibric Acid 105 mg Tablets | Fenofibrate 145 mg Tablets
Number analyzed (Participants) | 47 | 47
ng-hr/mL | 121,974.07 (46,243.60) | 132,463.37 (48,121.11)

3. Primary Outcome: The Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity AUC(0-∞)
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: Pharmacokinetic analyses are based on 47 out of 54 enrolled subjects who completed this study.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Fenofibric Acid 105 mg Tablets | Fenofibrate 145 mg Tablets
Number analyzed (Participants) | 47 | 47
ng-hr/mL | 134,576.33 (52,676.64) | 146,847.53 (54,588.94)

ADVERSE EVENTS:
Description: 54 subjects were enrolled in this study. Several subjects dropped out of the study prior to receiving both interventions. 51 subjects were administered Fenofibric Acid 105 mg tablets. 50 subjects were administered Fenofibrate 145 mg tablets.
Groups:
- Fenofibric Acid 105 mg Tablets: Each subject received one tablet of fenofibric acid 105 mg 30 minutes after the initiation of a standard breakfast.
- Fenofibrate 145 mg Tablets: Each subject received one tablet of fenofibrate 145 mg 30 minutes after the initiation of a standard breakfast.
Arm/Group | Fenofibric Acid 105 mg Tablets | Fenofibrate 145 mg Tablets
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 7/51 | 5/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibric Acid 105 mg Tablets (N=51) | Fenofibrate 145 mg Tablets (N=50)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days